CLINICAL TRIAL: NCT02433015
Title: Neurophysiological and Immunological Effects of the Transition From Combustible to Electronic Cigarettes
Acronym: ECIG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Collaborators: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2014-004-00
Record Dates: First submitted 2015-04-24; First posted 2015-05-04 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Tobacco Smoking; Nicotine Dependence
Keywords: Electronic Cigarette
MeSH Terms: conditions — Tobacco Smoking; Tobacco Use Disorder; Vaping | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tobacco Cigarette Group (Active Comparator): This group will not receive an electronic cigarette and will continue to smoke combustible tobacco cigarettes as previously.
  Interventions: Other: Tobacco Cigarette
- Electronic Cigarette Group (Experimental): This group will receive an electronic cigarette to use for the duration of the study.
  Interventions: Other: Electronic Cigarette

INTERVENTIONS:
Other: Electronic Cigarette — eGo-type electronic cigarette with a supply of 18mg/ml nicotine solution
  Arms: Electronic Cigarette Group
Other: Tobacco Cigarette — Smoke own brand of cigarette as previously
  Arms: Tobacco Cigarette Group

SUMMARY:
The objective of this study is to examine the cognitive, immunological, and neurophysiological effects of transitioning from tobacco cigarettes to electronic cigarettes. The central hypothesis of this study is that this transition will be accompanied by a decrease in peripheral inflammation, which will lead to significant changes in the neurocircuitry underlying interoception and appetite.

DETAILED DESCRIPTION:
Participants who are current cigarette smokers will be randomly assigned to either the experimental or control groups. Following a baseline psychiatric assessment session, subjects will return to the study center for two to three additional follow-up visits.

During the second visit, all subjects will undergo a functional magnetic resonance imaging (fMRI) scanning session, during which they will perform a series of functional neuroimaging tasks designed to examine the neural substrates involved in visceral interoception and eating behavior. Prior to the start of the scan session, blood samples will be collected from each subject, for the measurement of bio-markers related to nicotine use and peripheral inflammation. After the end of the second visit, subjects within the experimental group will be asked to switch from combustible to electronic cigarettes. Subjects within the control group will continue to smoke combustible cigarettes as previously.

During the third visit, which will follow two to eight weeks after the second visit, all subjects will provide a second blood sample and complete a second fMRI scan session. Both groups of participants will complete the same fMRI tasks as they did during the second visit.

ELIGIBILITY:
Inclusion Criteria:

* current cigarette smokers who have smoked for at least one year
* right-handed adults
* able to provide written informed consent

Exclusion Criteria:

* use of anticonvulsant, stimulant, or antipsychotic medication for 3 weeks prior to scanning
* any medical conditions or medications likely to influence cerebral blood flow or neurological function including cardiovascular, respiratory, endocrine and neurological diseases
* any history of drug (other than nicotine) or alcohol abuse within 1 year
* current pregnancy or breast feeding
* primary language other than English
* meeting general MRI exclusion criteria such as magnetic implants or claustrophobia
* Past history of any axis I psychiatric condition, other than major depressive disorder and post-traumatic stress disorder
* Current major depression or post-traumatic stress disorder
* Serious suicidal ideation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2015-01; Primary Completion 2016-09-24 (Actual); Study Completion 2016-09-24 (Actual)

PRIMARY OUTCOMES:
Change in overall levels of peripheral inflammatory cytokines | 2-8 weeks
  A composite measure of change in overall blood serum levels of multiple peripheral cytokines (CRP, TNF-alpha, sVCAM, IL-1RA, IL-6) between study visits two and three.

SECONDARY OUTCOMES:
Change in cotinine levels | 2-8 weeks
  Change in serum cotinine levels between study visits two and three.
Frequency of Electronic Cigarette use | 2-8 weeks
  Daily use of electronic cigarette between study visits two and three.
Change in exhaled Carbon Monoxide | 2-8 weeks
  Change in exhaled Carbon Monoxide between study visits two and three.
Frequency of Tobacco Cigarette use | 2-8 weeks
  Average number of tobacco cigarettes smoked between study visits two and three.
Change in Blood Oxygen Level-Dependent (BOLD) resting state functional connectivity during fMRI | 2-8 weeks
  Difference in resting-state functional connectivity between brain regions, measured by z-scores of correlated spontaneous fluctuations of the BOLD fMRI signal, between study visits two and three.
Change in BOLD fMRI response during interoception | 2-8 weeks
  Difference in the brain's hemodynamic response during a task of interoceptive attention to visceral signals, measured by percent change of the BOLD fMRI signal, between study visits two and three.
Change in BOLD fMRI response to food pictures | 2-8 weeks
  Difference in the brain's hemodynamic response to viewing pictures of appetizing food, measured by percent change of the BOLD fMRI signal, between study visits two and three.

CONTACTS AND LOCATIONS:
Overall Officials: William K Simmons, Ph.D, Principal Investigator — Laureate Institute for Brain Research
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States